CLINICAL TRIAL: NCT04540120
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of Orally Administered Dapansutrile Capsules for the Treatment of Moderate COVID-19 Symptoms and Evidence of Early Cytokine Release Syndrome
Brief Title: Safety and Efficacy of Dapansutrile for Treatment of Moderate COVID-19 Symptoms and Evidence of Early Cytokine Release Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to the treatment environment for COVID-19 evolving with the pervasiveness of vaccinations and other therapeutic modalities in mitigating against severe infection that has eliminated a viable patient population for study enrollment.
Sponsor: Olatec Therapeutics LLC (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OLT1177-10
Record Dates: First submitted 2020-08-13; First posted 2020-09-07 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Covid19; Cytokine Release Syndrome
Keywords: NLRP3; Covid19; Cytokine Release Syndrome; Dapansutrile
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — dapansutrile

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to receive either dapansutrile capsules or placebo capsules in a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a randomized, blinded, placebo-controlled study. Treatment allocation (to active or placebo treatment groups) will be blinded to all study participants, personnel, and investigators. Only the drug labeling personnel, unblinded pharmacist and DMC members may be unblinded to the treatment assignment. Also, in the event of an emergency, an unblinding envelope can be opened unmasking the treatment assignment to the PI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dapansutrile capsules (Experimental): Subjects will receive 4 x 250mg dapansutrile capsules BID for 14 days with an initial (first) dose of 8 x 250mg (2000 mg) administered at the study site on Day 1 (Day 1 dose may be 3000 mg).
  Interventions: Drug: dapansutrile capsules
- placebo capsules (Placebo Comparator): Subjects will receive 4 placebo capsules BID for 14 days with an initial (first) dose of 8 capsules administered at the study site on Day 1.
  Interventions: Drug: placebo capsules

INTERVENTIONS:
Drug: dapansutrile capsules — Hard opaque capsules containing 250 mg of API.
  Other Names: OLT1177 capsules
  Arms: dapansutrile capsules
Drug: placebo capsules — Hard opaque capsules containing 0 mg of API.
  Arms: placebo capsules

SUMMARY:
The purpose of this study is to assess the safety and efficacy of orally administered NLRP3 inhibitor, dapansutrile, for the treatment of moderate COVID-19 symptoms and early cytokine release syndrome (CRS) in patients with confirmed SARS-CoV-2 infection and moderate symptoms.

Coronavirus disease 2019 (COVID-19) is caused by infection from a new strain of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). COVID-19 is characterized by fever, cough and shortness of breath, which in certain patients can lead to systemic organ failure and mortality.

The data show that SARS-CoV-2 activates the innate immune signaling sensor NLRP3. Activation of NLRP3 initiates the cytokine release syndrome (CRS), which includes the production of primary cytokine, IL-1, triggering an intense inflammatory response that is prevalent in symptomatic COVID-19 patients. When CRS advances further to a fulminant 'cytokine storm', the data show that respiratory distress syndrome and multiple-organ failure take place.

A specific inhibitor of NLRP3, dapansutrile may reduce or prevent the hyperinflammation associated with CRS by inhibiting the production of IL-1β early to arrest the progression to a severe 'cytokine storm.' The end result would be a reduction in the need for COVID-19 patients to receive intensive medical treatment, allowing for fewer hospitalizations, administration of mechanical ventilation and deaths.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled study evaluating dapansutrile versus placebo. Approximately 80 subjects randomized 1:1 (40 dapansutrile, 40 placebo) are planned to be enrolled.

At the Screening/Baseline/Day 1 Visit, subjects will provide informed consent, be screened for eligibility, and be randomized/enrolled into the study. Subjects will also receive the first dose of study drug at this visit once study eligibility has been confirmed, and the second dose of study drug will be taken approximately 12 hours after the first dose. Study drug will be continued twice daily (morning and evening doses) through Day 14.

The trial duration will be approximately 45 days for all subjects enrolled, with assessments as follows: Screening/Baseline/Day 1, Day 4 (±1 day), Day 8 (±1 day), Day 15 (±1 day), Day 29 (±3 days), and Day 45 (± 3 days). The Day 29 and Day 45 follow-up visits will be conducted virtually via the institution's telehealth process.

Each subject will be asked to maintain two paper diaries at home daily for the first 14 days: a dosing diary and a subject diary. The dosing diary will be used to record the number of capsules taken each morning and evening. The subject diary will be used to record temperature, oxygen levels, COVID-19 symptoms, and overall health (using the prior 24-hour period for parameters requiring subject recall). The set of questions used in the subject diary will also be administered to the subjects at the Screening/Baseline/Day 1 Visit (pre-dose), Day 15, Day 29, and Day 45 visits. Each subject will be provided a no-contact thermometer and a hand-held pulse oximeter at the Screening/Baseline/Day 1 Visit for home use.

At Day 29 and Day 45, additional assessments of safety and clinical activity will occur. The Day 29 and Day 45 follow-up visits will be conducted virtually via the sites' telehealth process.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥ 18 years of age;
2. SARS-CoV-2-positive, confirmed by Food and Drug Administration (FDA)- or European Medicines Agency (EMA)-authorized COVID-19 test ≤ 7 days prior to randomization;
3. Less than or equal to 7 days from first symptom onset to randomization;
4. Subjects with moderate COVID-19 consistent with the definition of "moderate" as set forth by the February 2021 FDA Guidance for Industry: COVID-19: Developing Drugs and Biological Products for Treatment or

   Prevention (FDA, 2021) who at the Screening/Baseline/Day 1 Visit:
   1. have felt feverish within the past 24 hours,
   2. have an SpO2 > 93% on room air at sea level when sitting, and
   3. meet at least one of the following criteria: i). Respiratory rate: ≥ 20 breaths/minute, when the subject is sitting, ii). SpO2: ≤ 96% on room air at sea level, when the subject is sitting, iii). Shortness of breath: with exertion, not requiring oxygen, or vi). Heart rate: ≥ 90 beats/minute, when the subject is sitting;
5. If all the criteria in Inclusion 4c are met, subject must possess at least one of the following high-risk conditions known to have an underlying increased level of cytokine production; otherwise, at least two of these high-risk conditions must be met:

   1. 70 years or more of age,
   2. Obesity (BMI ≥ 30 kg/m2),
   3. Diabetes (type 1 or 2),
   4. Uncontrolled hypertension, defined as diastolic > 100 mm Hg and/or systolic > 150 mm Hg without any current anti-hypertensive medications. At the time of screening if the subject is on anti- hypertensive medication(s) and diastolic or systolic rates are elevated, subject may be enrolled after consultation with the Medical Monitor,
   5. Known respiratory disease (including asthma or chronic obstructive pulmonary disease [COPD]),
   6. Known heart failure (note: subjects with New York Heart Association Class IV congestive heart failure cannot be enrolled per Exclusion Criterion 4), or
   7. Known coronary disease;
6. Plasma CRP level must be collected at Screening/Baseline/Day 1 Visit;
7. Acceptable overall medical condition to be safely enrolled in and complete the study (with specific regard to cardiovascular, renal, and hepatic conditions) in the opinion of the Investigator;
8. Ability to provide written, informed consent prior to initiation of any study- related procedures, and ability in the opinion of the Investigator to understand and comply with all the requirements of the study, which includes abstaining from the use of prohibited medications.
9. Subject must present with at least moderate symptomatology, based on having symptoms in the prior 24 hours that were uncomfortable and interfered with daily activities or required treatment other than study drug and having at least one of the following symptoms: cough; fatigue; myalgia; diarrhea; vomiting; nausea; headache; sore throat; nasal congestion; rhinorrhea; loss of taste; loss of smell; fainting; or chills, shivering, and/or sweating.

Exclusion Criteria:

1. Women of childbearing potential, or men whose sexual partner(s) is a woman of childbearing potential, who:

   1. Are or intend to become pregnant (including use of fertility drugs) during the study;
   2. Are nursing (female subjects only);
   3. Are not using an acceptable, highly effective method of contraception until all follow-up procedures are complete.
2. Evidence of pre-existing or new-onset organ failure;
3. Evidence of moderate concurrent nervous system, renal, endocrine, or gastrointestinal disease, unrelated to COVID-19 as determined by the Investigator;
4. Evidence of cardiovascular disease with significant arrhythmia, congestive heart failure (New York Heart Association Class IV), unstable angina, cor pulmonale, or symptomatic pericardial effusion, not related to COVID-19 as determined by the Investigator;
5. Required use of vasoactive drug support;
6. History of myocardial infarction in the 6 months prior to the Screening/Baseline/Day 1 Visit;
7. Evidence of current liver disease, not related to COVID-19 as determined by the investigator;
8. History or evidence of active tuberculosis (TB) infection at Screening/Baseline/Day 1 Visit or one of the risk factors for tuberculosis such as but not limited or exclusive to:

   1. History of any of the following: residence in a congregate setting (e.g., jail or prison, homeless shelter, or chronic care facility), substance abuse (e.g., injection or non-injection), health-care workers with unprotected exposure to subjects who are at high risk of TB or subjects with TB disease before the identification and correct airborne precautions of the subject or
   2. Close contact (i.e., share the same air space in a household or other enclosed environment for a prolonged period (days or weeks, not minutes or hours)) with a person with active pulmonary TB disease within the last 12 months.
9. History of or currently active primary or secondary immunodeficiency;
10. Past or present requirement for oxygen (e.g., nasal cannula, proning, mechanical ventilation and/or supplemental oxygen).
11. Use of any prohibited concomitant medications/therapies over the defined or planned use of any concomitant medications/therapies during the

    Treatment Period, including specifically:
    1. use of ibuprofen or diclofenac
    2. use of colchicine
    3. use of systemic steroids within 30 days of randomization
    4. use of janus kinase (JAK) inhibitors
    5. use of off-label agents (e.g., hydroxychloroquine, remdesivir, dexamethasone) and biologic and oral anti-cytokine agents (e.g., current treatment with adalimumab, infliximab, etanercept, golimumab, certolizumab pegol, tocilizumab, sarilumab, anakinra, canakinumab, rilonacept, baricitinib, tofacitinib, or upadacitinib);

    Note: During the treatment period a patient may meet the criteria for a treatment approved by the FDA specifically for COVID-19 (e.g. remdesivir). In this situation the investigator and medical monitor should confer and take the most appropriate decision for the patient. If possible, the preference would be for the patient to complete the 14 days of dosing before adding on the 2nd treatment. If that is not possible the preference would be for the patient to continue their 14 days on dapansutrile and complete all study related visits.
12. Known history of renal impairment (e.g., calculated glomerular filtration rate [GFR] < 45 mL/min);
13. Evidence of malignant disease, or malignancies diagnosed within the previous 5 years (except for local basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured);
14. History of infection or known active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV);
15. Any other concomitant medical or psychiatric conditions, diseases, or prior surgeries that, in the opinion of the Investigator, would impair the subject from safely participating in the trial and/or completing protocol requirements;
16. Individuals who have been in a chronic care facility in the past 30 days;
17. Individuals who are incarcerated;
18. Participation in any clinical trial and/or use of any investigational product within the immediate 30-day period prior to the Screening/Baseline//Day 1 Visit; or receipt prior to Screening/Baseline/Day 1 Visit or intending to receive during the trial a COVID-19 vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with clinical deterioration | Day 15
  Clinical deterioration is defined as having any COVID-19-related hospitalization after enrollment or both (1) worsening or persistence of shortness of breath and (2) oxygen saturation less than 92% on room air at sea level or need for supplemental oxygen to achieve oxygen saturation of 92% or greater.

SECONDARY OUTCOMES:
Proportion of subjects with complete resolution of fever symptoms and shortness of breath | Day 8, Day 15, Day 29, Day 45
  Complete resolution is defined as having a symptom described as "absent" on the subject diary with no return of the symptom before Day 45.
Cumulative incidence of SAEs | Day 45
  Evaluate the cumulative incidence of SAEs of dapansutrile relative to placebo
Cumulative incidence of Grade 3 and Grade 4 Adverse Events | Day 45
  Evaluate the cumulative incidence of Grade 3 and Grade 4 Adverse Events of dapansutrile relative to placebo
Discontinuation or temporary suspension of participation | Day 45
  Evaluate the cumulative incidence of discontinuation or temporary suspension (for any reason) of dapansutrile relative to placebo
Changes in white cell count | Day 8, Day 15
  Evaluate changes in white cell count of dapansutrile relative to placebo over time
Changes in hemoglobin | Day 8, Day 15
  Evaluate changes in hemoglobin of dapansutrile relative to placebo over time
Changes in platelets | Day 8, Day 15
  Evaluate changes in platelets of dapansutrile relative to placebo over time
Changes in creatinine | Day 8, Day 15
  Evaluate changes in creatinine of dapansutrile relative to placebo over time
Changes in glucose | Day 8, Day 15
  Evaluate changes in glucose of dapansutrile relative to placebo over time
Changes in total bilirubin | Day 8, Day 15
  Evaluate changes in total bilirubin of dapansutrile relative to placebo over time
Changes in ALT | Day 8, Day 15
  Evaluate changes in ALT of dapansutrile relative to placebo over time
Changes in AST | Day 8, Day 15
  Evaluate changes in AST of dapansutrile relative to placebo over time
Incidence of new infection that occurs during the study | Day 8, Day 15
  Evaluate changes in incidence of new infection that occurs during the study of dapansutrile relative to placebo
Incidence of opportunistic infections | Day 8, Day 15
  Evaluate changes in incidence of opportunistic infections of dapansutrile relative to placebo
Time to clinical improvement | Baseline/Day 1 to Day 15
  Time to clinical improvement in fever symptoms and shortness of breath
Time to sustained absence of fever | Baseline/Day 1 to Day 15
  Time to sustained absence of fever, defined as at least 2 days since last temperature measurement of ≥ 38˚C (100.4°F)
Clinical improvement in symptoms relevant to COVID 19 | Day 15
  Proportion of subjects who experience clinical improvement in symptoms relevant to COVID 19 (e.g., cough, diarrhea, vomiting)
Incidence of hospitalization, supplemental oxygen, mechanical ventilation, or death before Day 15 | Day 15
  Incidence of subjects meeting the composite endpoint of subjects requiring hospitalization (hospitalization is defined as ≥ 24 hours of acute care), supplemental oxygen, mechanical ventilation, or who die
Duration of hospitalization, supplemental oxygen or mechanical ventilation before Day 15 | Day 15
  Duration of incidences of subjects meeting the composite endpoint of subjects requiring hospitalization (hospitalization is defined as ≥ 24 hours of acute care), supplemental oxygen or mechanical ventilation
Clinical improvement in symptoms | Baseline/Day 1 to Day 15
  Proportion of subjects who experience clinical improvement in symptoms by Day 15, defined as a reduction of two or more points on the WHO Ordinal Scale for Clinical Improvement (lowest score between Baseline Visit/Day 1 and Day 15)
Improvement in oxygenation | Baseline/Day 1 to Day 15
  Improvement in oxygenation over the course of the study and maintenance of this effect
Change in ALT | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in AST
Change in AST | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in AST
Change in blood glucose | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in blood glucose
Change in Erythrocyte Sedimentation Rate (ESR) | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in Erythrocyte Sedimentation Rate (ESR)
Change in Hemoglobin A1c (HbA1C) | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in Hemoglobin A1c (HbA1C)
Change in Lactate dehydrogenase (LDH) | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in Lactate dehydrogenase (LDH)
Change in Lymphocyte, Absolute count | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in Lymphocyte, Absolute count
Change in Monocyte, Absolute count | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in Monocyte, Absolute count
Change in Neutrophils, Absolute count | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in Neutrophils, Absolute count
Change in Eosinophil, Absolute count | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in Eosinophil, Absolute count
Change in CRP | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in CRP
Change in D-Dimer | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in D-Dimer
Change in Ferritin | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in Ferritin
Change in Fibrinogen | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in Fibrinogen
Change in Partial Thromboplastin Time (PTT) and International Normalized Ratio (INR) | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in Partial Thromboplastin Time (PTT) and International Normalized Ratio (INR)
Change in IL-1β | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in IL-1β
Change in IL-6 | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in IL-6
Change in IL-18 | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in IL-18
Change in granulocyte colony-stimulating factor (G-CSF) | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in granulocyte colony-stimulating factor (G-CSF)
Change in interferon-γ-induced protein 10 (IP-10) | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in interferon-γ-induced protein 10 (IP-10)
Change in C3a | Baseline/Day 1 to Day 15
  Assess and compare change from Baseline in C3a

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - C&R Research Services USA, Coral Gables, Florida
  - Invesclinic U.S. LLC, Fort Lauderdale, Florida
  - Inpatient Research Clinic, LLC, Hialeah, Florida
  - Sunrise Research Institute, Sunrise, Florida
  - Las Vegas Medical Research, LLC, Las Vegas, Nevada
  - PanAmerican Clinical Research LLC, Brownsville, Texas
  - J & S Studies, Inc., College Station, Texas
  - C&R Research Services USA, Houston, Texas
  - Texas Research Alliance LLC, McAllen, Texas
- University Hospital Basel, Basel, Switzerland